CLINICAL TRIAL: NCT06986343
Title: Effect of Palatal Expansion and Up-Locker Activator on Sleep Architecture and Pharynx Dimensions in Children
Brief Title: Impact of Palatal Expansion and Up-Locker Activator on Sleep and Pharyngeal Dimensions in Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Claudia Cecilia Restrepo Serna, PhD. Director CES-LPH Research Group, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CES1198
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Breathing Disorder During Sleeping; Sleep Habits
Keywords: Palatal expansion; Up-Locker vacuum activator; polysmonography; airway; Hyrax; Children
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind, randomized controlled clinical trial will be performed. Children aged 6 to 8 years, recruited from the clinics of the postgraduate program of Pediatric Dentistry and the private practice of one of the investigators (CR), will be included. The sample size was calculated based on the differences reported by Sökücü et al. Assuming a 95% confidence level, 80% power, and a 20% treatment difference, 17 participants per group (total n = 34) will be required. No additional oversampling will be planned due to ethical considerations regarding radiation exposure.
  The inclusion criteria will include the presence of sleep-disordered breathing symptoms with a minimum score of 6 on the Spanish version of the Children's Sleep Habits Questionnaire (CSHQ), documented snoring recorded by RONCOLAB® for at least five consecutive days, and transverse maxillary deficiency of at least 5 mm, defined as a superior intermolar distance of le
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1. Hyrax (Active Comparator): Children in the control group will have treatment with a semi-rapid maxillary expansion (SRME) with a Hyrax device with a Leone™ standard expansion screw. Bands will be placed on the maxillary first permanent molars, and a frame containing the maxillary canines and primary first molars will be used to support the expander. The same expert technician will construct all expanders. In both groups, the expander screw will be activated a quarter turn twice a day for the first 7 days, then once a day until the palatal cusp of the upper molar comes into contact with the buccal cusp of the lower molar. After the active phase, the expanders will be maintained in the oral cavity for 4 months for retention.
  Interventions: Device: Hyrax
- Group 2. Hyrax + Uplocker vacuum activator (Experimental): The patients in the intervention group (Hyrax+Up-locker vacuum activator) will receive a standardized training device (Up-Locker Vacuum Activator from Forwardontics™, approved by the FDA) immediately after finishing the retention period and retiring the expansion Hyrax device. Following instruction, the patients will undergo 30 minutes of daily home training in the first week, 60 minutes of daily home training in the second and third weeks, and thereafter 120 minutes of daily home training until completion of a 90-day program.
  Interventions: Device: Hyrax and Uplocker Vacuum Device

INTERVENTIONS:
Device: Hyrax — Children in this group are going to use only the Hyrax device.
  Arms: Group 1. Hyrax
Device: Hyrax and Uplocker Vacuum Device — Children in this group are going to use the Hyrax device and Up-Locker vacuum activator.
  Arms: Group 2. Hyrax + Uplocker vacuum activator

SUMMARY:
Objective: The study will aim to compare the effect of palatal expansion with Hyrax and Hyrax combined with Up-Locker on sleep behavior, sleep architecture, quality of life and nasal and pharyngeal airway dimensions, as well as intermolar, intercanine, and palatal depth dimensions in children. Materials and Methods: This prospective, single-blind, randomized controlled clinical trial will enroll 34 children aged 6-8 years, who will be randomly assigned to receive treatment with either the Hyrax expansion appliance alone or in combination with the Up-Locker vacuum activator. Intercanine, intermolar, and palatal depth dimensions will be evaluated through intraoral scans. Airway dimensions will be assessed using panoramic and lateral cephalometric radiographs, while sleep behavior will be analyzed with the Children's Sleep Habits Questionnaire (CSHQ) and sleep architecture will be evaluated via polysomnography. Data will be analyzed using the Shapiro-Wilks test for homogeneity, and comparisons will be performed with either the t-test or the Mann-Whitney U test. Results: It is expected that intercanine and intermolar distances will improve in both the Hyrax and Hyrax combined with Up-Locker vacuum activator groups after treatment, while palatal depth will present a significant reduction only in the group receiving Hyrax with Up-Locker. The group using the Hyrax combined with Up-Locker vacuum activator will likely experience more significant improvements in sleep latency, total sleep time, REM sleep, and arousal indices compared to the Hyrax group (p<0.05) after treatment. Both groups are anticipated to demonstrate reduction of snoring, enhanced airway dimensions post-treatment, including the area of the nostrils and the naso and oropharynx. Conclusion: It is expected that combined treatment with Hyrax and Up-Locker vacuum activator will yield superior outcomes in sleep architecture, intraoral dimensions, and airway dimensions.

DETAILED DESCRIPTION:
This investigation was approved by the ethics committee of Universidad CES, and the parents will provide their written informed consent while the children will give their written assent. A prospective, single-blind, randomized controlled clinical trial will be performed. Children aged 6 to 8 years will be recruited from the clinics of the postgraduate program of Pediatric Dentistry and the private practice of one of the investigators (CR).

The sample size will be calculated based on the differences reported by Sökücü et al., assuming a 95% confidence level, 80% power, and a 20% treatment difference. According to the analysis, 17 participants per group (total n = 34) will be required.

Snoring will be recorded using SnoreLab®, a validated mobile application created to monitor and analyze snoring behavior, providing insights into sleep patterns and potential underlying sleep disorders. Utilizing advanced sound detection technology, the app will record snoring episodes during the night, delivering detailed feedback on the frequency and intensity of snoring. Users will need to demonstrate valid recordings for at least 50% of each night. Data collection will continue until five nights of recordings are achieved. To be included in the study, participants will be required to exhibit snoring-whether light, loud, or epic-across these five nights.

Weight will be measured at the Universidad CES clinic or the private practice of one of the investigators (CR), using a standard physician's scale, ensuring that the children will be dressed in light clothing and not wearing shoes. The scale will provide a precision of 0.1 kg. Height will be assessed using a wall-mounted height board, adhering to the following criteria: children will stand barefoot, with heels together, and with their heels, buttocks, shoulders, and head in contact with the wall while maintaining a neutral gaze. Measurements will be recorded to the nearest 0.1 cm. BMI will then be calculated using the formula kg/m².

Participants will be randomly assigned using a random number generator with REDCap® to one of two groups: Group 1 - Control group (Treatment with the Hyrax expansion appliance alone) or Group 2 - Intervention (Treatment with the Hyrax appliance in combination with the Up-Locker vacuum activator).

Intervention For both groups, the semi-rapid maxillary expansion (SRME) will be performed using a Hyrax device with a Leone™ standard expansion screw in all children. Bands on the maxillary first permanent molars and a frame containing the maxillary canines and primary first molars will be used to support the expander. All expanders will be constructed by the same expert technician. In both groups, the expander screw will be activated a one-quarter turn twice a day for the first 7 days, then once a day until the palatal cusp of the upper molar comes into contact with the buccal cusp of the lower molar. After the active phase, the expanders will be maintained in the oral cavity for 4 months as retention.

Patients in Group 2 will receive a standardized training device (Up-Locker Vacuum Activator from Forwardontics™, approved by the FDA) immediately after finishing the retention period and retiring the expansion Hyrax device. The patients will be instructed to gather saliva while positioning the Up-locker vacuum activator between their front teeth and lips, using a mirror to monitor the placement of the membrane within the funnel. During the swallowing of saliva, negative pressure formation will be observed with the Up-locker vacuum activator by inversion of the membrane into the funnel. The patients will be informed that the goal of the treatment is to establish a nasal breathing pattern and a tongue resting posture against the palate to help stabilize both the tongue and the soft palate. They will be advised to refrain from creating excessive negative pressure during the exercises to prevent any adverse effects related to pressure on the gums. Following instruction, the patients will undergo 30-minute daily home training the first week, 60-minute daily home training the second and third weeks, and afterwards 120-minute daily home training until the completion of a 90-day program. The recommendation will be to use the afternoon, while watching TV or reading, or in the evening before rest. Revisions of adequate use of the device will be performed by the investigator (CR) every 4 weeks.

Outcome Measures Sleep behavior Sleep behavior will be assessed with the validated CSHQ, which is a 35-item questionnaire administered to parents, asking them to report their child's sleep behaviors and patterns during the last typical week. The questionnaire will be developed to address significant clinical sleep complaints commonly observed in this age group and will provide data on the following subscales (with score ranges in parentheses): Bedtime Resistance (6-36), Sleep Onset Delay (1-3), Sleep Duration (3-9), Sleep Anxiety (4-12), Night Awakenings (3-9), Parasomnias (7-21), Sleep Disordered Breathing (3-9), Daytime Sleepiness (8-24). Each item on the questionnaire will be rated on a three-point scale: "usually" (5-7 times a week) = 3, "sometimes" (2-4 times a week) = 2, and "rarely" (0-1 time a week) = 1. A composite score will be computed as the sum of scores on the 33 items across all subscales. A total score of 41 will be considered the clinical cut-off, indicating a potential risk of sleep problems.

Sleep architecture All children in the control and intervention group will undergo a one-night PSG study in a sleep laboratory in Medellín, Colombia, before treatment (T0) and at the end of treatment of the intervention group (T1, nine months after the beginning of treatment for both groups). The sleep study will use a sleep recording system and dedicated scoring software (Neuron-Spectrum-65/PSG system™, Neurosoft Ltd. Ivanova, Russia). The measurements will be taken between 9:00 pm and 6:00 am for all participants. Audio and video signals will be captured in parallel. A nasal flow cannula and a thermistor respiratory monitor will record the respiration, and a finger pulse oximeter will monitor blood oxygen saturation (SaO2). A trained research team will install all electrodes and sensors.

The sleep architecture will be evaluated according to the AASM Manual for the Scoring of Sleep and Associated Events. The following measures will be taken:

* Total sleep duration (TSD): cumulative time (in hours) spent in non-REM (nREM) stages 1, 2, and 3 and Rapid Eye Movement (REM) sleep from sleep onset to lights-on time.
* Sleep onset latency (SOL): elapsed time between light-out time and the first occurrence of any sleep stage other than a stage of awakening.
* Time and proportion spent in each sleep stage: cumulative time and proportion of sleep spent in each sleep stage (nREM stages 1, 2, and 3 (N3 and N4 will be grouped) and REM sleep) between sleep onset and lights-on time.
* Arousals/hour during REM and nREM sleep: 3-5 seconds of arousal (abrupt alterations of oscillatory patterns, characterized by low-voltage fast-rhythm EEG oscillations during REM and nREM sleep).

ELIGIBILITY:
Inclusion Criteria:

* The Inclusion Criteria will include the presence of sleep-disordered breathing symptoms with a minimum score of 6 on the Children's Sleep Habits Questionnaire (CSHQ), documented snoring recorded by SnoreLab® for at least five consecutive days, and transverse maxillary deficiency of at least 5 mm, with a normal superior intermolar distance defined as a minimum of 40 mm (measured between the mesiopalatine cusps of teeth 16 and 26).

Exclusion Criteria:

* The exclusion criteria for this study will include a history of previous treatment for OSA (including tonsillectomy and adenoidectomy), being overweight or obese (Body Mass Index (BMI) at or above the 85th percentile for their age and sex), chronic systemic diseases unrelated to upper airway respiratory alterations (e.g., chronic cardiopulmonary or neuromuscular diseases), facial malformations (e.g., syndromes with facial or cleft lip/palate anomalies, or clinically evident palatal malformations), presence of dental caries, previous treatment with maxillary orthopedics or orthodontics, and failure to comply with scheduled control visits.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Sleep behavior | From enrollment to the end of treatment at 9 months
  Sleep behavior will be assessed using the validated CSHQ, which is a 35-item questionnaire that will be administered to parents, asking them to report their child's sleep behaviors and patterns during the last typical week. The questionnaire will be developed to address significant clinical sleep complaints commonly observed in this age group and will provide data on the following subscales (with score ranges in parentheses): Bedtime Resistance (6-36), Sleep Onset Delay (1-3), Sleep Duration (3-9), Sleep Anxiety (4-12), Night Awakenings (3-9), Parasomnias (7-21), Sleep Disordered Breathing (3-9), and Daytime Sleepiness (8-24). Each item on the questionnaire will be rated on a three-point scale: "usually" (5-7 times a week) = 3, "sometimes" (2-4 times a week) = 2, and "rarely" (0-1 time a week) = 1. A composite score will be computed as the sum of scores on the 33 items across all subscales.
Sleep architecture | From baseline to the end of treatment at 9 months
  Sleep architecture would be assessed with polysomnography All children in the control and the intervention group will undergo a one-night PSG study in a sleep laboratory in Medellín, Colombia, before treatment (T0) and at the end of treatment for the intervention group (T1, nine months after the beginning of treatment for both groups). The sleep study will utilize a sleep recording system and dedicated scoring software (Neuron-Spectrum-65/PSG system™, Neurosoft Ltd. Ivanova, Russia). The measurements will be made between 9:00 pm and 6:00 am for all participants. Audio and video signals will be recorded in parallel. A nasal flow cannula and a thermistor respiratory monitor will record respiration, and a finger pulse oximeter will monitor blood oxygen saturation (SaO2). A trained research team will install all electrodes and sensors.
  The sleep architecture will be evaluated according to the AASM Manual for the Scoring of Sleep and Associated Events.
Pharynx dimensions | From baseline to the end of treatment at 9 months
  Dimensions of the naropharynx and oropharynx are going to be measured in lateral cephalic x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia C Restrepo-Serna, PhD, Principal Investigator — CES University
Locations (1):
- Dentistry Faculty, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The laws regarding the protection of personal data and research in Colombia (from which the research subjects will be selected) are quite strict when it comes to children. Therefore, the database of participants will only be shared upon request from external researchers, and after a careful assessment of the reasons for the request.

REFERENCES:
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Dutil C, Walsh JJ, Featherstone RB, Gunnell KE, Tremblay MS, Gruber R, Weiss SK, Cote KA, Sampson M, Chaput JP. Influence of sleep on developing brain functions and structures in children and adolescents: A systematic review. Sleep Med Rev. 2018 Dec;42:184-201. doi: 10.1016/j.smrv.2018.08.003. Epub 2018 Aug 15. PMID 30241996
- [Derived] Restrepo C, Kahn S, Gozal D. Impact of Palatal Expansion With Up-Locker on Children With Sleep-Disordered-Breathing: A Clinical Trial. Pediatr Pulmonol. 2026 Jan;61(1):e71424. doi: 10.1002/ppul.71424. PMID 41521856

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT06986343/Prot_SAP_ICF_000.pdf